CLINICAL TRIAL: NCT02391194
Title: A Phase 1 Trial of AVB-620 in Women With Primary, Non-Recurrent Breast Cancer Undergoing Surgery
Brief Title: Trial of AVB-620 in Women With Primary, Non-Recurrent Breast Cancer Undergoing Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avelas Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVB620-C-001
Record Dates: First submitted 2015-02-20; First posted 2015-03-18 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: AVB-620; stage I; newly diagnosed; breast cancer; stage II; stage III; ductal carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVB-620 (Experimental): Eligible subjects will receive a single dose of AVB-620 as an intravenous infusion before the surgical procedure.
  Interventions: Drug: AVB-620

INTERVENTIONS:
Drug: AVB-620

SUMMARY:
This is a Phase 1, open-label, dose escalation study in women with primary, non-recurrent breast cancer undergoing surgery. AVB-620 will be administered prior to surgery.

DETAILED DESCRIPTION:
This study will examine the safety and tolerability of AVB-620 administered as an IV infusion to women with primary, non-recurrent breast cancer undergoing surgery. The study will also characterize the pharmacokinetics of AVB-620 in this subject population and determine the dose of AVB-620 needed to generate a fluorescence signal in tumor and lymph node tissue to enable fluorescence recordings and image analysis with an imaging system. The study will also evaluate the effect of timing of AVB-620 administration, relative to surgery, on fluorescence characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Ductal carcinoma in situ (DCIS) or Stage I-III, primary invasive carcinoma of the breast
* Primary surgical treatment is planned to be a mastectomy or lumpectomy. Sentinel lymph node (LN) biopsy or axillary LN dissection (ALND) is planned as part of the subject's therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate renal function
* Lab values (hematology and chemistry) within institution's normal laboratory limits
* Willing to remain on-site for approximately 24 hours after administration of AVB-620 or, if required, stay overnight after the surgical procedure
* If the subject received neoadjuvant therapy, residual tumor is present (to be determined by the primary surgeon)
* If the subject received prior anthracycline therapy, the left ventricular ejection fraction (LVEF) must be within institution's normal limits
* Subject has the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Recurrent ipsilateral breast cancer
* Prior neoadjuvant chemotherapy or biologic therapy for current clinically or biopsy-proven node positive breast cancer within 4 weeks before the planned surgery.
* Open surgery in the ipsilateral breast within 1 year of AVB-620 administration
* History of radiation therapy to ipsilateral breast
* Abnormal cardiac rhythm not controlled with medication, history of stroke, coronary events, and/or heart failure within 1 year of AVB-620 administration
* Diagnosis of autoimmune disorders
* History of drug-related anaphylactic reactions or allergic reactions; subjects with an active diagnosis of uncontrolled airway hyperactivity, uncontrolled asthma, or asthma requiring oral corticosteroids will be excluded
* History of renal disease or current evidence of renal disease
* Current diagnosis of any other active or clinically significant non-breast cancer
* Systemic investigational drug of any kind within 6 weeks of AVB-620 administration
* Pregnant or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Safety of AVB-620 as assessed by the incidence of adverse events and abnormal laboratory values | 30 days
  The incidence, nature and severity of adverse events and abnormal laboratory values will be collected and analyzed in the evaluation of the safety of AVB-620.

SECONDARY OUTCOMES:
Characterize the pharmacokinetic profile of AVB-620 | 8 days
  The pharmacokinetics (PK) of AVB-620 will be characterized by collecting and reviewing individual subject plasma concentrations and primary parameters, including clearance, Cmax, Cmin, and distribution.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Moores UC San Diego Cancer Center, La Jolla, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Hospitals and Clinics, Stanford, California